CLINICAL TRIAL: NCT07142889
Title: The Effectiveness of Blood Flow Restriction Training on Patellar Position, Muscle Morphology, and Lower Limb Function in Patients After Anterior Cruciate Ligament Reconstruction
Brief Title: BFR Training for Post ACLR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, I Putu Gde Surya Adhitya, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1937/UN14.2.2.VII.14/LT/2025
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Blood Flow Restriction Training; Patella Position; Muscle Morphology; Anterior Cruciate Ligament Reconstruction; Leg Function

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low load-BFRt (Experimental): 70% of the arterial occlusion pressure and 30% of the maximum repetition rate
  Interventions: Procedure: Low load-BFRt
- Sham Low load-BFRt (Sham Comparator): 10% of the arterial occlusion pressure and 30% of the maximum repetition rate
  Interventions: Procedure: Sham Low load-BFRt
- High load-Eccentric training (Active Comparator): 70% of the maximum repetition rate
  Interventions: Procedure: High load-Eccentric training

INTERVENTIONS:
Procedure: Low load-BFRt — The participants' two legs will be subjected to 70% arterial occlusion pressure when the physical therapist applies the BFR cuffs. After that, participants will be required to complete eccentric exercises with a maximum repetition count of 30%, such as single leg squat, single leg deadlift, lateral step down, dan single leg calf raise.
  Arms: Low load-BFRt
Procedure: Sham Low load-BFRt — The participants' two legs will be subjected to 10% arterial occlusion pressure when the physical therapist applies the BFR cuffs. After that, participants will be required to complete eccentric exercises with a maximum repetition count of 30%, such as single leg squat, single leg deadlift, lateral step down, dan single leg calf raise.
  Arms: Sham Low load-BFRt
Procedure: High load-Eccentric training — The physical therapist will instruct the participants to complete eccentric exercises at a maximum of 70% repetitions, such as single leg squat, single leg deadlift, lateral step down, dan single leg calf raise.
  Arms: High load-Eccentric training

SUMMARY:
This randomized clinical trial is designed to compare three different rehabilitation methods for patients who have undergone anterior cruciate ligament (ACL) reconstruction. The study aims to determine whether low-load blood flow restriction training (LL-BFRt) is more effective than high-load eccentric training (HL-Et) and a sham LL-BFRt in improving three key areas: patellar position, muscle morphology, and leg function.

Study Design and Interventions

Participants will be randomly assigned to one of the three intervention groups. All groups will perform eccentric exercises, including single leg squats, single leg deadlifts, lateral step downs, and single leg calf raises. The key differences lie in the load and the use of blood flow restriction:

LL-BFRt Group: Participants will train at 30% of their repetition maximum (RM) while a cuff restricts blood flow to 70% of their artery occlusion pressure (AOP).

HL-Et Group: Participants will train at a higher intensity, using 70% of their repetition maximum (RM), with no blood flow restriction.

Sham LL-BFRt Group: Participants will perform the same exercises as the LL-BFRt group at 30% of their RM, but the cuff will not be inflated to a pressure that restricts blood flow.

After the training period, the researchers will compare the outcomes across all three groups to see which method leads to the most significant improvements in patella position, muscle morphology, and leg function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15-35 years old.
* History of a unilateral ACL injury, underwent ACL reconstruction surgery more than 6 months ago, and completed rehabilitation with physiotherapy.
* Adults participating in recreational or competitive sports at a minimum of level 3 on the Tegner Activity Scale.
* No prior history of a grade 3 sprain/strain injury to other tissues in the knee and foot.
* No recurring knee injuries after the ACL reconstruction surgery.
* Willing to be a research subject from start to finish by signing an informed consent form.

Exclusion Criteria:

* Hypertension, circulatory disorders, sickle cell anemia, obesity, diabetes, kidney disorders, venous thromboembolism, cancer, and tumors are contraindications for BFR application.
* Experiencing a disability or being disabled.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Patella position | 8 weeks
  Using a musculoskeletal ultrasonography, researchers will determine the patella position.
Muscle cross-sectional area | 8 weeks
  Using a musculoskeletal ultrasonography, researchers will determine the cross-sectional area of vastus medial obliques muscle and hamstring muscles.
Vastus medial obliques fiber angle | 8 weeks
  Using a musculoskeletal ultrasonography, researchers will determine the vastus medial obliques fiber angle.
Quadriceps strength | 8 weeks
  Using a hand-held dynamometer, researchers will determine the isometric quadriceps muscle.
Dynamic balance | 8 weeks
  Using a modified star excursion balance test, researchers will determine the distance of three positions of legs reaching, including forward, posteromedial, and posterolateral.
Leg function | 8 weeks
  Using KOOS questionnaires will determine the subjective score of the patient's leg function.
Anterior knee pain | 8 weeks
  Using the Kujala questionnaire will determine the subjective score of the patient's knee pain levels.

SECONDARY OUTCOMES:
Incidence of anterior cruciate ligament reinjury | 1 year
  Researchers will determine the incidence of anterior cruciate ligament reinjury with the physical examination of Lachman's test.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical therapy laboratory, College of Medicine, Universitas Udayana and ROM Physiotherapy Private Clinic Denpasar, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No